CLINICAL TRIAL: NCT01304043
Title: Observatoire Francophone Des Tumeurs Malignes Rares de l'Ovaire : Protocole de Prise en Charge Chez l'Adulte (Tumeurs Germinales et Des Cordons Sexuels)
Brief Title: French Observatory of Rare Malignant Tumors of the Ovary
Status: Completed | Type: Observational
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Other Study IDs: TMRO
Record Dates: First submitted 2005-09-09; First posted 2011-02-25 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Ovarian Tumors
Keywords: ovarian tumors; rare ovarian tumors; germinal tumors; sexual cords tumors; observatory; forum
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: chemotherapies protocols — Cisplatine 20 mg/m² IV Etoposide 100 mg/m² IV Bléomycine 30 mg IV

SUMMARY:
To take charge of the treatment in rare adult ovarian tumors with an homogenous manner (germinal and sexual cords tumors), at different stages of the disease.

DETAILED DESCRIPTION:
* to establish prognosis factors for the disease
* to proceed in a centralised examination of histologic laminas
* to reach in the long-term and homogenous follow-up of the patients
* to follow-up the long-term toxicities of the treatments given
* to analyse and follow-up the later fertility of the patients
* to evaluate the interest of setting a multi-disciplinary discussion forum on the Web

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* germinal or sexual cords ovary tumors histologically proven
* first line or relapse treatment
* written informed consent

Exclusion Criteria:

* mental ineptitude to understand and follow the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female with rare ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2002-01; Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Ray-Coquard, Physician, Principal Investigator — GINECO
Locations (1):
- Oncologie, Hôtel-Dieu, 1 place du parvis Notre-Dame, Paris, France

REFERENCES:
- See also: information for patients, discussion forum about "difficult" cases, therapeutic strategy for patients presenting rare ovarian tumor — http://www.ovaire-rare.org